CLINICAL TRIAL: NCT06949267
Title: A Prospective, Randomized Controlled Study of Human Induced Pluripotent Stem Cell-derived Mesenchymal Stromal Cells (iMSC) for the Prevention of Acute Graft-versus-host Disease After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: A Study of iMSC for the Prevention of Acute Graft-versus-host Disease After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RJ-BMT-GvHD-001
Record Dates: First submitted 2025-03-26; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Acute Graft-versus-Host Disease
Keywords: iMSC; III-IV aGVHD; allogeneic hematopoietic stem cell transplantation; prophylaxis

STUDY DESIGN:
Intervention Model Description: enrolled subjects will be 1:1 randomly assigned to experimental group or control group.The control group will receive conventional aGVHD prophylaxis and the experimental group will be receive iMSC injection plus the conventional aGVHD prophylaxis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): conventional aGVHD prophylaxis
  Interventions: Combination Product: conventional aGVHD prophylaxis
- Trial group (Experimental): conventional aGVHD prophylaxis + iMSC
  Interventions: Biological: iMSC; Combination Product: conventional aGVHD prophylaxis

INTERVENTIONS:
Biological: iMSC — 1× 10^6/kg each time, twice a week
  Arms: Trial group
Combination Product: conventional aGVHD prophylaxis — Cyclosporine or tacrolimus(CNI)+Mycophenolate mofetil(MMF)± Short Course Methotrexate(MTX)+Anti-human T-lymphocyte Globulin（ATG）

SUMMARY:
An open-label, randomized, controlled clinical trial to explore the efficacy and safety of iMSC in preventing the development of acute graft-versus-host disease of degree III-IV in patients after allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
This is an open-label, randomized, controlled study, enrolled subjects(patients at risk for aGVHD of degree III-IV after allogeneic hematopoietic stem cell transplantation) will be 1:1 randomized to experimental group or control group. Control group will receive conventional aGVHD prophylaxis and the experimental group will receive iMSC injection plus conventional aGVHD prophylaxis, with 28 cases in each group, for a total of 56 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with malignant or nonmalignant hematologic diseases 7-21 days after allogeneic hematopoietic stem cell transplantation;
* No gender restrictions and age between 14-70 years old；
* Patients received aGVHD prophylaxis regimen of a calcium-modulated phosphatase inhibitor combined with mycophenolate mofetil wtih or without short-course methotrexate and rabbit anti-human thymocyte globulin (CNI+MMF± short-course MTX +ATG)；
* Patients had a MAGIC algorithm probability (MAP) score ≥ 0.14 at +7d or +14d after allogeneic hematopoietic stem cell transplantation(HSCT) (if patients had a MAP< 0.14 at +7d, another test was performed at +14d)；
* Estimated survival≥ 24 weeks；
* Eastern Cooperative Oncology Group（ECOG）≤ 2 points and Hematopoietic Cell Transplantation Comorbidity Index (HCT-CI)≤ 3 points；
* Subjects were be treated within 5 days after enrollment；
* Informed consent and willingness to participate in the study.

Exclusion Criteria:

* Serious organ dysfunction such as organ failure after allogeneic HSCT;
* Received more than once HSCT (including autologous transplants);
* Positive for Hepatitis B Surface Antigen (HBsAg) or Hepatitis B Core Antibody (HBcAb) and have Hepatitis B Virus (HBV) DNA titers above the normal range ; positive for Hepatitis C Virus (HCV) antibodies and have positive peripheral blood HCV RNA; positive for Human Immunodeficiency Virus (HIV) antibodies; positive for syphilis;
* Subjects with severe hepatic veno-occlusive disease or sinus veno-occlusive syndrome;
* Primary malignant hematologic disease was not remission;
* Within 6 months prior to enrollment, subjects had other diseases or their physiological conditions may interfere the study results, or had life-threatening complications;
* Those who are suffering mental or neurological illnesses, unable to express will correctly;
* Those with active malignant solid tumors within 5 years prior to participation in this study, with the exception of radically treated cervical cancer, in situ limited prostate cancer, and nonmelanoma skin cancer;
* Subjects known to be potentially allergic or highly sensitized to the cell therapy in the study protocol;
* Have participated or are participating in another clinical trial within one month prior to enrollment;
* Those who are judged by the investigator to be unsuitable for participation in this clinical trial.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of degree III-IV aGvHD | Within 100 days of first dose
  Cumulative incidence of degree III-IV aGvHD at 100 days Within 100 days of first dose

SECONDARY OUTCOMES:
Cumulative Recurrence Rate (CIR) | Day 100, Month 6, Month 9, Month 12 , Month 18 , Month 24 after first dose
  Cumulative Recurrence Rate (CIR) at Day 100, Month 6, Month 9, Month 12 , Month 18 , Month 24 after first dose
Disease-free survival (DFS) | Day 100, Month 6, Month 9, Month 12 , Month 18 , Month 24 after first dose
  DFS at Day 100, Month 6, Month 9, Month 12 , Month 18 , Month 24 after first dose
Adverse Event(AE) or Serious Adverse Event(SAE) | Day 100 after initial infusion
  Number of participants with treatment-related adverse events or serious adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxia Hu, MD, Principal Investigator — Ruijin Hospital